CLINICAL TRIAL: NCT06075264
Title: A Phase II Double-blind, Placebo-controlled, Randomized Trial of Topical Artesunate Ointment for the Treatment of Patients With Vulvar High-grade Squamous Intraepithelial Lesions (Vulvar HSIL)
Brief Title: Phase II Study of Artesunate Ointment for the Treatment of Vulvar High Grade Squamous Intraepithelial Lesions (Vulvar HSIL, VIN2/3)
Acronym: ART-VIN IIB
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Frantz Viral Therapeutics, LLC (Industry)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ART-VIN IIB; 23-889 (Other: Cleveland Clinic IRB)
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Vulvar Diseases; HPV Infection; Vulvar HSIL; Pre-Cancerous Dysplasia; HPV Disease; VIN, Usual Type; VIN 2 of Usual Type; VIN 3 of Usual Type; Vin II; Vin III; VIN Grade 2; VIN Grade 3; High Grade Intraepithelial Neoplasia
Keywords: topical treatment; ointment; non-surgical; vulvar cancer prevention; high-risk HPV; human papillomavirus; HPV; vulvar HSIL; High grade lesions
MeSH Terms: conditions — Vulvar Diseases; Papillomavirus Infections | interventions — artesunic acid; artenimol; artemisinin

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled randomized trial
Who Masked: Participant, Investigator
Masking Description: Double-blind, placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Artesunate ointment (Active Comparator): Artesunate formulated as topical ointment, 40% Four 5-day cycles of artesunate ointment every 2 weeks
  Interventions: Drug: Artesunate ointment
- Placebo ointment (Placebo Comparator): Placebo ointment Four 5-day cycles of placebo ointment every 2 weeks
  Interventions: Drug: Placebo ointment

INTERVENTIONS:
Drug: Artesunate ointment — topical ointment, as a non-surgical treatment
  Other Names: Artesunic acid; Dihydroartemisinin (DHA); Artemisinin
  Arms: Artesunate ointment
Drug: Placebo ointment — topical placebo ointment
  Other Names: Placebo to artesunate ointment
  Arms: Placebo ointment

SUMMARY:
This is a phase II double-blind, placebo-controlled study of artesunate ointment for the treatment of HPV-associated vulvar HSIL (usual type vulvar intraepithelial neoplasia 2/3).

DETAILED DESCRIPTION:
Eligible participants in this study are randomized 2:1 to receive either artesunate or placebo ointment for the treatment of vulvar HSIL. Both groups receive four 5-day cycles of topical ointment, at weeks 0, 2, 4, and 6. Dosing visits may be done in person or as telehealth (ointment may be shipped directly to the patient). Participants are followed closely with vulvar examinations or colposcopies at weeks 8, 18, 6-months and 12-months.

ELIGIBILITY:
Inclusion Criteria:

* Adult women age ≥ 18 years
* Capable of informed consent
* Able to collaborate with planned follow-up (transportation, compliance history, etc)
* Biopsy diagnosis of high-grade vulvar dysplasia (VIN2, VIN3, VIN2/3, HSIL), including both new and recurrent disease. A biopsy diagnosis of vulvar high-grade squamous intraepithelial lesion within the previous 3 months which was not excised or otherwise treated may be accepted for study entry.
* Positive HPV test at study entry (any genotype).
* Women of childbearing potential agree to use birth control during the dosing phase (through week 8).
* Laboratory values at Screening of:

  * Serum alanine transaminase (SGPT/ALT) < 5 x upper limit of normal (ULN)
  * Serum aspartate transaminase (SGOT/AST) < 5 x ULN
  * Serum Bilirubin (total) < 2.5 x ULN
  * Serum Creatinine ≤ 1.5 x ULN
* Weight ≥ 50kg

Exclusion Criteria:

* Pregnant and nursing women
* Concurrent anal, vulvar, or cervical cancer
* HIV-positive participants with a CD4 count < 200
* Participants infected with HIV-1 if not on a stable, suppressive antiretroviral therapy (ART) regimen.
* Unwillingness to undergo an excisional procedure at week 18 to either remove HSIL lesions, or to document histologic regression at a site where HSIL was present at study entry.
* Currently receiving systemic chemotherapy or radiation therapy for another cancer.
* Concomitant use of Efavirenz for HIV antiretroviral treatment
* Concomitant use of strong UGT inhibitors
* Concomitant use of imiquimod, cidofovir, or 5-fluorouracil (5-FU) for the duration of the study
* Concurrent dermatological conditions affecting the vulva (e.g., herpetic lesion, Crohn's disease, hidradenitis suppurativa) or vulvar dermatoses (e.g., lichen sclerosis or planus, atopic dermatitis, genital atrophy).
* Concurrent treatment with systemic corticosteroids

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is only for biological females
Enrollment: 27 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with complete histologic response | 18 weeks
  Number of participants who have complete histologic response following topical artesunate ointment

SECONDARY OUTCOMES:
Number of participants who have achieved viral clearance | Week 18
  Number of participants who achieve clearance of HPV genotypes present at screening. These genotypes become undetectable over the study window.
Number of participants who show partial response | Week 18
  Number of participants with documented partial response following topical artesunate
Number of participants who have durable response | Week 18
  Number of participants with documented complete response who do not have recurrence of their vulvar HSIL over the study window
Incidence of Treatment-Emergent Adverse Events (TEAE) | 8 weeks
  Number of participants who report artesunate-related serious adverse events

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Florida Gynecologic Oncology, Fort Myers, Florida
  - Ascension St. Vincent, Indianapolis, Indiana
  - Cleveland Clinic Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Hillcrest Hospital, Mayfield Heights, Ohio

IPD SHARING:
Plan to Share IPD: No